CLINICAL TRIAL: NCT01648348
Title: Phase I/Comparative Randomized Phase II Trial of TRC105 Plus Bevacizumab Versus Bevacizumab in Bevacizumab-Naive Patients With Recurrent Glioblastoma Multiforme
Brief Title: Bevacizumab With or Without Anti-Endoglin Monoclonal Antibody TRC105 in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01989; NCI-2012-01989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000737109; N1174; NCCTG-N1174; N1174 (Other: Alliance for Clinical Trials in Oncology); N1174 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — carotuximab; Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (bevacizumab and TRC105) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 and 11 of course 1 and days 1 and 8 of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-Endoglin Chimeric Monoclonal Antibody TRC105; Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment
- Arm II (bevacizumab) (Active Comparator): Patients receive bevacizumab as in arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Anti-Endoglin Chimeric Monoclonal Antibody TRC105 — Given IV
  Other Names: TRC105
  Arms: Arm I (bevacizumab and TRC105)
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar FKB238; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This partially randomized phase I/II trial studies the side effects and the best dose of anti-endoglin monoclonal antibody TRC105 when given together with bevacizumab and to see how well they work in treating patients with glioblastoma multiforme that has come back. Monoclonal antibodies, such as anti-endoglin monoclonal antibody TRC105 and bevacizumab, may find tumor cells and help kill them. Giving anti-endoglin monoclonal antibody TRC105 together with bevacizumab may be an effective treatment for glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a maximum tolerated dose (MTD) of TRC105 (anti-endoglin monoclonal antibody TRC105) combined with bevacizumab in this patient population. (Phase I) II. To assess the safety and adverse events of TRC105 in combination with bevacizumab in this patient population. (Phase II) III. To determine the efficacy of TRC105 in combination with bevacizumab in recurrent glioblastoma as measured by progression-free survival and compare it with the efficacy of bevacizumab alone in this patient population. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the proportion of patients, who are progression free at 6 months, treated with TRC105 in combination with bevacizumab as compared to bevacizumab alone. (Phase II) II. To assess the overall survival of patients treated with TRC105 in combination with bevacizumab compared to bevacizumab alone. (Phase II) III. To compare the impact of the treatment on the patients quality of life (QOL) using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ)-C15-Palliative Care (PAL) and QLQ-brain neoplasm (BN)20 Patient Questionnaires. (Phase II) IV. To estimate patient recommendations for study participation to others using the Was It Worth It (WIWI) Questionnaire. (Phase II)

TERTIARY OBJECTIVES:

I. To evaluate the pharmacokinetics of TRC105. (Phase I) II. To evaluate the immunogenicity of TRC105. (Phase I) III. To determine the relationship between tumor biomarkers, circulating biomarkers of vascular response and vascular endothelial growth factor (VEGF)/VEGF receptor (VEGFR) single-nucleotide polymorphisms (SNPs) in predicting efficacy and/or toxicity of treatment. (Phase II) IV. To assess the utility of magnetic resonance imaging (MRI) imaging including apparent diffusion coefficient (ADC) as a predictor of response and survival. (Phase II) V. To assess the utility of dynamic contrast enhanced (DCE) MRI as a predictor of response to bevacizumab with or without TRC105. (Phase II)

OUTLINE: This is a phase I dose-escalation study of anti-endoglin monoclonal antibody TRC105, followed by a randomized phase II study.

Phase I (closed to accrual 1/14/14): Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 and 11 of course 1 and days 1 and 8 of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Phase II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 and 11 of course 1 and days 1 and 8 of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab as in arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of grade 3 or 4 glioma, including astrocytoma, oligodendroglioma, and mixed gliomas, as determined by pre-registration central pathology review (Phase I)
* Histological confirmation of glioblastoma multiforme (grade 4 astrocytoma) as determined by pre-registration central pathology review; note: gliosarcomas and other grade 4 astrocytoma variants (e.g., giant cell) are eligible; glioblastoma (GBM) with oligodendroglial features are NOT PERMITTED in this study if they are 1p19q co-deleted; sites submitting GBM with oligodendroglial features will be asked to provide results of 1p/19q co-deletion status (Phase II)
* Evidence of tumor progression by MRI or computed tomography (CT) scan following radiation therapy or following the most recent anti-tumor therapy; note: patients who have had surgical treatment at recurrence are eligible if they had a resection with measurable or non-measurable residual disease on postoperative imaging or if there is imaging evidence of disease progression as compared to the first postoperative scan
* Measurable or evaluable disease by gadolinium MRI or contrast CT scan; note: patients who have had a gross total resection (GTR) are eligible on the basis of evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* White blood cells (WBC) >= 3,000/mL
* Hemoglobin >= 10.0 g/dL; note: this level may be reached by transfusion
* Total bilirubin =< institutional upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2 x ULN
* Creatinine =< ULN
* Life expectancy >= 12 weeks
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Urine protein creatinine (UPC) ratio < 1; note: urine protein must be screened by urine analysis for UPC ratio; for UPC ratio >= 1.0, 24-hour urine protein must be obtained and the level should be < 1,000 mg for registration
* Fixed or decreasing dose of corticosteroids (or no corticosteroids) >= 7 days prior to registration
* Calculated glomerular filtration rate (GFR) must be >= 60 ml/min; GFR will be calculated as needed per institutional guidelines
* Any number of prior chemotherapy regimens for recurrent disease (Phase I); =< 1 chemotherapy or other non-antiangiogenic regimen for recurrent disease (Phase II)
* Last dose of bevacizumab >= 2 weeks prior to registration (Phase I); note: for the phase II study only, prior exposure to bevacizumab is not allowed
* Surgery >= 4 weeks prior to registration
* Completion of radiation therapy >= 12 weeks prior to registration and prior chemotherapy >= 4 weeks prior to registration (>= 6 weeks from nitrosourea-containing regimens)
* Small molecular cell cycle inhibitors >= 2 weeks from registration
* Ability to provide informed written consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willing to return to enrolling institution for follow-up
* Willing to discontinue use of medications that inhibit platelet function >= 10 days prior to registration; aspirin at doses greater than 325 mg/day must be discontinued >= 10 days prior to registration and avoided through the study; note: nonsteroidal anti-inflammatory drug (NSAID) medications are recommended in place of aspirin; if NSAIDs or aspirin are used, histamine (H)-2 blockers and proton pump inhibitor (PPI) medications are recommended
* Willing to provide mandatory blood and tissue samples for correlative research purposes (Phase I and II)

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the duration of the study and for at least 6 months after treatment has ended
* Prior hypersensitivity to bevacizumab or toxicity requiring discontinuation of bevacizumab (Phase I)
* Any prior exposure to any VEGF or VEGF inhibitor including, but not limited to, bevacizumab, cediranib, vandetanib, sunitinib, pazopanib, aflibercept, or sorafenib (Phase II)
* Prior hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies (Phase I and II)
* Prior hypersensitivity to triptan derivatives (Phase I and II)
* Other active malignancy =< 3 years prior to registration; exceptions: non-melanotic skin cancer or carcinoma-in-situ of the cervix; note: if there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* Uncontrolled infection
* Immunocompromised patients or patients known to be human immunodeficiency virus (HIV) positive and currently receiving combination antiretroviral therapy; patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* History of hypertensive crisis or hypertensive encephalopathy
* Clinically significant cardiovascular disease defined as follows:

  * Inadequately controlled hypertension (i.e., systolic blood pressure [SBP] > 160 mm Hg and/or diastolic blood pressure [DBP] > 90 mm Hg despite antihypertensive therapy)
  * History of cerebrovascular accident (CVA) within 6 months
  * Myocardial infarction or unstable angina within 6 months
  * New York Heart Association classification II, III, or IV cardiovascular disease
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (i.e., aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* Evidence or history of bleeding diathesis (greater than normal risk of bleeding, i.e., hereditary hemorrhagic telangiectasia type I or HHT-1) or coagulopathy in the absence of therapeutic anti-coagulation or any hemorrhage/bleeding event > grade 3 within 4 weeks prior to registration; note: patients with full-dose anticoagulants are eligible provided the patient has been on a stable dose for at least 2 weeks of low molecular weight heparin; therapeutic Coumadin and aspirin doses > 325 mg daily are not allowed
* Receiving any other investigational agent that would be considered as a treatment for the primary neoplasm
* Prior treatment with TRC105
* Serious or non-healing wound, active ulcer, or untreated bone fracture
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 6 months prior to registration
* History of invasive procedures defined as follows:

  * Major surgical procedure, open biopsy, or significant traumatic injury =< 28 days prior to registration
  * Anticipation of need for major surgical procedures during the study
  * Core biopsy =< 7 days prior to registration
* History of significant vascular disease (i.e., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) within 6 months prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05-11 (Actual); Study Completion 2017-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (308):
- United States (308):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Saint Jude Medical Center, Fullerton, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Maine Center for Cancer Medicine-Scarborough, Scarborough, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Ann Arbor Hematology -Oncology Associates, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OneHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University Medical Center Brackenridge, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Bev + TRC105 (Dose 0, Cohort A): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 (as 3 mg/kg IV) and 11 (as 3 mg/kg IV) of course 1 and days 1 (as 6 mg/kg IV)and 8 (as 6 mg/kg IV) of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I: Bev + TRC105 (Dose 1, Cohort A): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 (as 3 mg/kg IV) and 11 (as 5 mg/kg IV) of course 1 and days 1 (as 8 mg/kg IV)and 8 (as 8 mg/kg IV) of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I: Bev + TRC105 (Dose 2, Cohort A); Phase I: Bev + TRC105 (Dose 2, Cohort B): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 (as 3 mg/kg IV) and 11 (as 7 mg/kg IV) of course 1 and days 1 (as 10 mg/kg IV)and 8 (as 10 mg/kg IV) of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase II: Bev + TRC105 (Arm I): Experimental: Arm I (bevacizumab and TRC105): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on day 1 and 10 mg/kg anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 and 11 of course 1 and days 1 and 8 of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase II: Bev Alone (Arm II): Active Comparator: Arm II (bevacizumab): Patients receive bevacizumab as in arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I: Bev + TRC105 (Dose 0, Cohort A) | Phase I: Bev + TRC105 (Dose 1, Cohort A) | Phase I: Bev + TRC105 (Dose 2, Cohort A) | Phase I: Bev + TRC105 (Dose 2, Cohort B) | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Started | 5 | 3 | 4 | 3 | 52 | 49
Completed | 3 | 3 | 3 | 3 | 49 | 43
Not Completed | 2 | 0 | 1 | 0 | 3 | 6
Not completed — Cancel | 1 | 0 | 0 | 0 | 3 | 6
Not completed — Replaced for MTD analysis | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Bev + TRC105 (Dose 0-2): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 (as 3 mg/kg IV) and 11 (as 3/5/7 mg/kg IV) of course 1 and days 1 (as 6/8/10 mg/kg IV)and 8 (as 6/8/10 mg/kg IV) of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase I: Bev + TRC105 (Dose 0-2) | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II) | Total
Number analyzed (Participants) | 15 | 52 | 49 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (6.6) | 56.8 (12.3) | 55.6 (10.2) | 55.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 17 | 12 | 33
  Male | 11 | 35 | 37 | 83
Region of Enrollment [Number; unit: participants]
  United States | 15 | 52 | 49 | 116

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I) as Measured by the Number of Participants With Dose Limiting Toxicities
Description: MTD for this study will be defined as the highest safely tolerated dose level where at most 1 out of 6 patients experience dose-limiting toxicity (DLT) with the next higher dose having at least 2 patients out of a maximum of 6 patients experience DLT. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD. The number of DLT's will be reported here.
Time Frame: 28 days
Population: All phase I patients who completed the study were eligible and analyzed for MTD.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Bev + TRC105 (Dose 2, Cohort A + B): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on day 1 and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 8 (as 3 mg/kg IV) and 11 (as 7 mg/kg IV) of course 1 and days 1 (as 10 mg/kg IV)and 8 (as 10 mg/kg IV) of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I: Bev + TRC105 (Dose 0, Cohort A) | Phase I: Bev + TRC105 (Dose 1, Cohort A) | Phase I: Bev + TRC105 (Dose 2, Cohort A + B)
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 1

2. Primary Outcome: Progression-free Survival (PFS) (Phase II)
Description: Progression Free Survival time is defined as the time from study randomization to documentation of disease progression. Patients who die without documentation of progression will be considered to have had tumor progression at the time of death. Patients who fail to return for evaluation after beginning therapy will be censored for progression on the last day of therapy or date last known to be alive, whichever is later. Patients who are still alive and have not progressed will be censored for progression at the time of the last tumor assessment. The time-to-progression distribution will be estimated using the Kaplan-Meier method.
Time Frame: The time from study randomization to documentation of disease progression, assessed up to 2 years
Population: All phase II patients who started the study were eligible and analyzed for the primary outcome of Phase II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 52 | 49
months | 2.9 [2.8 to 4.9] | 3.2 [2.6 to 4.6]
Statistical Analysis 1: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Test type: Superiority; p = 0.57, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.73 to 1.77]

3. Secondary Outcome: Overall Toxicity Rate for Grade 3 or Higher Adverse Events Considered at Least Possibly Related to Treatment (Phase II)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment will be compared using a Fisher's Exact test between the 2 treatment groups.
Time Frame: Up to 2 years
Population: All phase II patients who completed the study were eligible and included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 49 | 43
percentage of patients | 57.1 | 16.3
Statistical Analysis 1: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Test type: Superiority; p < 0.001, Fisher Exact

4. Secondary Outcome: Overall Survival (Phase II)
Description: Survival time is defined to be the length of time from start of study therapy to death due to any cause. All patients meeting the eligibility criteria that have signed a consent form and begun treatment will be considered evaluable for estimation of the survival distribution. The distribution of overall survival for both groups of the study will be estimated using the Kaplan-Meier method, and be compared using log-rank tests.
Time Frame: The time from start of study therapy to death due to any cause, assessed up to 2 years
Population: All phase II patients who started the study were eligible and included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 52 | 49
months | 9.7 [6.7 to 11.5] | 7.4 [6.5 to 12.7]
Statistical Analysis 1: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Test type: Superiority; p = 0.82, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.66 to 1.69]

5. Secondary Outcome: Progression Free Survival at 6 Months (PFS6) (Phase II) as Measured by the Percentage of Participants With Progression Free Survival at 6 Months
Description: PFS6 is defined as the time from start of study therapy to the date of first observation of disease progression or death due to any cause (whichever comes first). The medians and confidence intervals given are the Kaplan-Meier estimates.
Time Frame: The time from study randomization to documentation of disease progression, assessed at 6 months
Population: All phase II patients who started the study were eligible and included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of progression-free patients
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 52 | 49
percentage of progression-free patients | 25.0 [15.3 to 40.8] | 30.2 [18.8 to 48.4]

6. Secondary Outcome: Quality of Life (QOL) as Assessed by the EORTC QLQ-C15-PAL Questionnaire [Item 15: Global Health Status/Quality of Life] (Phase II)
Description: Quality of Life (QOL) as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C15-PAL questionnaire, as measured by the change from baseline to the end of cycle 2 (4 weeks) in the EORTC QLQ-C15-PAL item 15, Global health status/quality of life, score. The assessment was scored using EORTC's scoring algorithms. The score range is from 0-100 (0 corresponding to worst outcome; 100 corresponding to best outcome). Range of the change in scores from baseline to cycle 2 (4 weeks) is (-100,100). The mean change in score and 95% confidence interval of the change from baseline to the end of cycle 2 (4 weeks) are reported below.
Time Frame: Baseline and 4 weeks
Population: All phase II patients who completed the EORTC QLQ-C15-PAL questionnaire at baseline and at the end of cycle 2 were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 35 | 30
units on a scale | -3.3 [-9.7 to 3.0] | 4.4 [-5.8 to 14.6]
Statistical Analysis 1: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Test type: Superiority; p = 0.19, t-test, 2 sided

7. Secondary Outcome: QOL Assessed by EORTC-QLQ-BN20 Patient Questionnaire [Items 1-20] (Phase II)
Description: QOL assessed by EORTC-QLQ-BN20 Patient Questionnaire (Brain cancer module), as measured by the change from baseline to the end of cycle 2 (4 weeks) in the EORTC QLQ-BN20 Items 1-20 are used to score the following 11 symptom scales: Future uncertainty (Items 1-3,5), Visual disorder (Items 6-8), Motor dysfunction (Items 10,15, 19), Communication deficit (Items 11-13), Headaches (Item 4), Seizures (Item 9), Drowsiness (Item 14), Itchy Skin (Item 17), Hair Loss (Item 16), Weakness of legs (Item 18), and Bladder control (Item 20). The assessment was scored using EORTC's scoring algorithms. The score range for each of the 11 symptom scales is from 0-100 (0 corresponding to not severe;100 corresponding to most severe). Range of changes in scores from baseline to cycle 2 (4 weeks) is (-100,100). The mean change in score and 95% confidence interval of each symptom scale are reported below.
Time Frame: Baseline and 4 weeks
Population: All phase II patients who completed the EORTC-QLQ-BN20 patient questionnaire at baseline and at the end of cycle 2 were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 36 | 30
units on a scale
  Future uncertainty | -8.0 [-15.3 to -0.7] | -11.9 [-23.0 to -0.9]
  Visual disorder | 2.0 [-1.7 to 5.7] | 5.9 [1.7 to 10.1]
  Motor dysfunction | 3.4 [-3.1 to 9.9] | 3.3 [-3.8 to 10.5]
  Communication deficit | 0.3 [-6.3 to 6.9] | 1.9 [-5.6 to 9.3]
  Headaches | 7.4 [-1.2 to 16.0] | 0 [-6.5 to 6.5]
  Seizures | -1.9 [-4.5 to 0.8] | -2.2 [-7.8 to 3.4]
  Drowsiness | 2.8 [-5.0 to 10.6] | 4.4 [-8.1 to 17.0]
  Itchy skin | -9.3 [-18.4 to -0.1] | -1.1 [-8.0 to 5.8]
  Hair loss | -0.9 [-7.2 to 5.4] | -2.2 [-8.7 to 4.3]
  Weakness of legs | 10.2 [0.9 to 19.5] | -2.2 [-14.4 to 10.0]
  Bladder control | 5.6 [-1.8 to 12.9] | 3.3 [-3.5 to 10.2]
Statistical Analysis 1: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Future uncertainty symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.55, t-test, 2 sided
Statistical Analysis 2: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Visual disorder symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.16, t-test, 2 sided
Statistical Analysis 3: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Motor dysfunction symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.99, t-test, 2 sided
Statistical Analysis 4: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Communication deficit symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.75, t-test, 2 sided
Statistical Analysis 5: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Headaches symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.17, t-test, 2 sided
Statistical Analysis 6: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Seizures symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.90, t-test, 2 sided
Statistical Analysis 7: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Drowsiness symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.82, t-test, 2 sided
Statistical Analysis 8: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Itchy skin symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.15, t-test, 2 sided
Statistical Analysis 9: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Hair loss symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.77, t-test, 2 sided
Statistical Analysis 10: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Weakness of legs symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 11: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Bladder control symptom scale/item t-test, 2-sided, unpooled; Test type: Superiority; p = 0.65, t-test, 2 sided

8. Secondary Outcome: QOL Assessed by WIWI Questionnaire (Phase II)
Description: Quality of life (QOL) assessed by Was it worth it? (WIWI) questionnaire, as measured by the percentage of patients answering yes to the question "Was it worthwhile for you to participate in this research study?"
Time Frame: Up to 4 weeks
Population: All phase II patients who completed the WIWI questionnaire were included in this analysis.
Measure: Number; unit: percentage of patients answering yes
Arm/Group | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
Number analyzed (Participants) | 36 | 32
percentage of patients answering yes | 69.4 | 71.9
Statistical Analysis 1: Comparison: Phase II: Bev + TRC105 (Arm I) vs Phase II: Bev Alone (Arm II); Test type: Superiority; p = 0.83, proportion test

9. Other Pre Specified Outcome: Change in DCE-MRI Utility
Description: Associations between the change of DCE-MRI and PFS6 will be assessed using two-sample t-test.
Time Frame: Baseline to up to 2 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in MRI ADC Utility
Description: MRI ADC histogram metrics such as overall ADC, mean ADC of lower curve, percentage of ADC in lower curve, and skewness at baseline and change from baseline to the first follow-up MRI will be analyzed for association with progression free and overall survival. Kaplan-Meier survival curves, logrank and Cox regression tests will be used to estimate and compare the equality of the overall survival and progression-time distributions of patient subsets defined by the ADC histogram metrics.
Time Frame: Baseline to up to 2 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Tumor and Circulating Biomarkers
Description: Binary endpoints and categorical endpoints will be compared using Chi-Squared or Fisher's Exact tests between treatment groups. Continuous endpoints will be analyzed using change-from-baseline measures and compared using t-tests between treatment groups and time-points. Cox proportional hazards regression will be used to determine if there are differences in PFS and OS between the treatment groups after correcting for each biomarker in conjunction with standard clinical variables.
Time Frame: Baseline to up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Description: The revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All graded AEs are reported. Cancels in the Participant Flow table did not receive treatment. Serious AE (SAE) reports for this study may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited Adverse Events (EAEs), and appear in the SAE table.
Arm/Group | Phase I: Bev + TRC105 (Dose 0, Cohort A) | Phase I: Bev + TRC105 (Dose 1, Cohort A) | Phase I: Bev + TRC105 (Dose 2, Cohort A) | Phase I: Bev + TRC105 (Dose 2, Cohort B) | Phase II: Bev + TRC105 (Arm I) | Phase II: Bev Alone (Arm II)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 2/49 | 2/43
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/3 | 1/4 | 2/3 | 15/49 | 8/43
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 3/3 | 48/49 | 38/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Bev + TRC105 (Dose 0, Cohort A) (N=4) | Phase I: Bev + TRC105 (Dose 1, Cohort A) (N=3) | Phase I: Bev + TRC105 (Dose 2, Cohort A) (N=4) | Phase I: Bev + TRC105 (Dose 2, Cohort B) (N=3) | Phase II: Bev + TRC105 (Arm I) (N=49) | Phase II: Bev Alone (Arm II) (N=43)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Bev + TRC105 (Dose 0, Cohort A) (N=4) | Phase I: Bev + TRC105 (Dose 1, Cohort A) (N=3) | Phase I: Bev + TRC105 (Dose 2, Cohort A) (N=4) | Phase I: Bev + TRC105 (Dose 2, Cohort B) (N=3) | Phase II: Bev + TRC105 (Arm I) (N=49) | Phase II: Bev Alone (Arm II) (N=43)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 2 (33) | 3 (25) | 36 (263) | 15 (38)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 1 (1) | 2 (12) | 2 (21) | 17 (86) | 11 (39)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (3) | 2 (4) | 13 (37) | 6 (14)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (22) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 5 (24) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (17) | 2 (35) | 0 (0) | 8 (12) | 7 (27)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (21) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (16) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (8) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (17) | 2 (11)
Fatigue (General disorders) | 3 (11) | 3 (21) | 3 (40) | 3 (18) | 44 (260) | 30 (254)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 2 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 11 (12) | 2 (2)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 6 (18) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 6 (7) | 5 (13)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 4 (7)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 14 (47) | 19 (81)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (19)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 8 (22) | 11 (58)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (9) | 3 (24)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (6) | 1 (5) | 9 (27) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (16) | 3 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (26)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (16) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (17) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (2)
Headache (Nervous system disorders) | 3 (7) | 3 (20) | 3 (37) | 3 (17) | 31 (158) | 16 (117)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 2 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 0 (0)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (13) | 3 (22)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (15) | 11 (22)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (8) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 13 (40) | 6 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (10) | 2 (30) | 2 (17) | 22 (141) | 4 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (20) | 1 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Body odor (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (16) | 1 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (20) | 0 (0) | 2 (10) | 2 (23)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (32) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (11) | 0 (0) | 0 (0) | 8 (17) | 4 (13)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 3 (37) | 1 (5) | 22 (136) | 28 (178)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less